CLINICAL TRIAL: NCT01439698
Title: Radio Frequency Ablation in the Management of Pancreatico-biliary Disorders: A Multicenter Registry
Acronym: RFA-Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Michel Kahaleh, Chief, Advanced Endoscopy, Weill Medical College of Cornell University
Other Study IDs: 1108011875
Record Dates: First submitted 2011-09-20; First posted 2011-09-23 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Cholangiocarcinoma; Pancreatic Cancer; Bile Duct Cancer; Biliary Stricture; Bile Duct Obstruction
Keywords: Cholangiocarcinoma; Pancreatic Cancer; Bile Duct Cancer; Biliary Stricture; Bile duct obstruction; ENDOHPB; Radio Frequency Ablation; RFA; ERCP; Endoscopic Retrograde Cholangiopancreatography; Registry; Multicenter
MeSH Terms: conditions — Cholangiocarcinoma; Pancreatic Neoplasms; Bile Duct Neoplasms; Cholestasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RFA for Pancreatico-biliary disorders: Subjects who will receive radiofrequency ablation for pancreatico-biliary disorders, including malignancies.
  Interventions: Device: Radio Frequency ablation Probe

INTERVENTIONS:
Device: Radio Frequency ablation Probe — Any probe that can conduct radiofrequency ablation within biliary ducts.
  Other Names: ENDOHPB

SUMMARY:
The objective of this protocol is to establish a multicenter registry to evaluate the impact of radiofrequency ablation in the management of patients with pancreatico-biliary disorders including malignancies.

DETAILED DESCRIPTION:
Bile duct cancer and pancreatic cancer are cancers that cannot be surgically removed. As the cancer grows, it blocks the drainage of the bile ducts that carry digestive juices from the gall bladder and pancreas to the small intestine. ERCP (endoscopic retrograde cholangiopancreatography) is often prescribed during which a tube with a tiny camera attached is inserted through the subject's mouth and advanced to a place in the small intestine where the bile duct empties. Through this scope the doctor enlarges the ducts with tiny balloons and places plastic or metal stents (straws) that help keep the bile ducts open so they can drain properly. However, due to the cancer, the stents are blocked eventually.

The purpose of this registry is to record information and evaluate the impact of radiofrequency ablation (RFA) of endoscopic radiofrequency ablation (RFA) probes in improving the management of bile duct cancer or pancreatic cancer by ablating the tissue in the bile duct(s) before the stent(s) are implanted. By using radiofrequency (RF) energy to heat the tissue in the duct(s) prior to stent(s) insertion, the surrounding tissue becomes coagulated and this may delay tumor growth and the time before the stent lumen becomes blocked. Thereby, allowing increased periods between the need for intervention and further stent implantation(s). The registry will evaluate the efficacy and safety of RFA procedures conducted for pancreatico-biliary disorders.

The safety and efficacy of various radio frequency ablation probes have been assessed in a series of studies. This multi-center registry has been initiated:

1. To document the immediate and post procedure clinical performance of radio frequency ablation in a 'real world' patient population requiring stent implantation for pancreaticobiliary disorders.
2. To assess the immediate and 6 months post procedure adverse event rate in patients.
3. To assess the impact of RFA on the life expectancy of patients suffering from pancreaticobiliary malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone RFA for pancreaticobiliary disorders
* Above 18 years of age

Exclusion Criteria:

* Patients who have not undergone RFA
* Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects over the age of 18 and suffering from pancreaticobiliary disorders, including malignancies such as Cholangiocarcinoma and Pancreatic Cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-09; Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Bile Duct Stricture Diameter. | 4 years
  Efficacy Assessment- Change from Baseline in Bile Duct Stricture Diameter.
Number of Participants with Adverse Events | 4 years
  Safety Assessment - Number of Participants with Adverse Events, type, frequency and intensity.

SECONDARY OUTCOMES:
Number of days of survival post intervention | 4 years
  Documentation of response rates,overall survival duration and overall stent occlusion-free duration.
Number of overall stent occlusion-free days post intervention | 4 years
  Documentation of overall stent occlusion-free duration post intervention to highlight quality of life and reduction of interventional procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York

IPD SHARING:
Plan to Share IPD: No
No IPD Sharing

REFERENCES:
- [Result] Sharaiha RZ, Natov N, Glockenberg KS, Widmer J, Gaidhane M, Kahaleh M. Comparison of metal stenting with radiofrequency ablation versus stenting alone for treating malignant biliary strictures: is there an added benefit? Dig Dis Sci. 2014 Dec;59(12):3099-102. doi: 10.1007/s10620-014-3264-6. Epub 2014 Jul 18. PMID 25033929